CLINICAL TRIAL: NCT05909592
Title: Epidemiological Profile and Shoulder Injury Risk Factors Investigation Among CrossFit Participants. Predictive Modeling for Shoulder Injury Incidence in These Populations.
Brief Title: Epidemiological Analysis of Shoulder Injuries Among Greek CrossFit Participants and Predictive Modeling for Shoulder Injury Incidence.
Status: Completed | Type: Observational
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Akrivi Bakaraki, Principal Investigator, University of Patras
Other Study IDs: 14279
Record Dates: First submitted 2023-05-01; First posted 2023-06-18 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Sports Injury; Shoulder Injuries; Risk Factors; Injury Prediction; Machine Learning; CrossFit
Keywords: Sports Injury; Shoulder Injuries; Risk Factors; Injury Prevention; Injury Prediction; Machine Learning; CrossFit
MeSH Terms: conditions — Athletic Injuries; Shoulder Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy CrossFit participants and athletes: No intervention. The group will be monitored for incidence data of shoulder injuries (new or aggravated pre-existing)

SUMMARY:
CrossFit is a modern sport, introduced to the public in 2000 and popular quickly with more than 15,000 affiliates worldwide. Due to the highly demanding nature of the workouts, it is claimed to be a sport with a high prevalence of injuries. Most preliminary retrospective studies had shown that shoulder area is injured most frequently, at about a quarter of all injuries. Therefore, the initial goal of this observational (prospective cohort) study is to learn about the incidence rates of shoulder injuries and potential risk factors in a Greek population of CrossFit participants. Based on these results, this study's ultimate purpose is to create a short warm-up program capable of reducing shoulder injuries and evaluate its effectiveness.

The main questions it aims to answer are:

* Are shoulder injuries as frequent as previous studies have shown to be?
* Can we blame for these injuries a previous history of musculoskeletal injury or deficits of range of motion, strength, and muscular endurance?
* Can a short warm up which targets revealed deficiencies be effective in reducing shoulder injuries incidence rates?

Participants will be asked to:

* take part in baseline measurements (personal data, previous musculoskeletal history, shoulder and core range of motion, shoulder and hip muscle strength, shoulder stabilizers endurance, functional assessment sport-specific tests)
* be monitored for new shoulder injuries or aggravation of old shoulder injuries that will occur during 12 months following baseline measurements. In this case, they must refer it to their coaches to be contacted and assessed by the researcher.
* be in touch with the researcher throughout the observational study and provide any required data regarding their participation

DETAILED DESCRIPTION:
CrossFit is prescribed as "a constantly varied, high-intensity, functional movement". It is a highly motivational way of training including a wide variety of different exercises modalities, including calisthenics, gymnastics, metabolic conditioning, and weightlifting, which includes both Olympic and powerlifting movements. This training model has been demonstrated to improve 10 physical skills: cardiovascular and respiratory endurance, stamina, strength, flexibility, power, speed, coordination, agility, balance, and accuracy. Its popularity has increased in recent years with more than 200,000 athletes competing worldwide and many more participants of a lower level. These characteristics led to concerns about CrossFit's safety, accordingly many researchers began to investigate whether the injury incidence rates are higher than other sports with retrospective studies, which were conducted via online questionnaires. The purpose of this prospective cohort study is to investigate shoulder injury rate among CrossFit participants in Greece and to design and examine the efficacy of a sport-specific injury prevention program in these kinds of injuries.

One hundred and eleven CrossFit participants will be surveyed. After reading and signing informed consent form, they will be interviewed for personal data, previous injuries history and general health. Shoulders and core range of motion, shoulders and hips muscle strength, shoulder stabilizers endurance will be measured with valid and reliable instruments. Also, functional assessment will be carry out using a novel instrument which has been developed in previous stage via a pilot study. CrossFit Screening Tool had been designed as a functional assessment instrument and applied as a pilot study to 20 CrossFit athletes. Based on the results, we have selected the functional tasks which will implement the baseline measurements process.

The sample will be monitored for any shoulder injury by the researcher for the following 12 months. In the term of shoulder injury is included any new or aggravated old injury which costs the athlete's absence or urges performance modifications for tissue protection. When an injury occurs, the researcher will contact the athlete, assess him using special questionnaires and clinical examination, including valid and reliable special clinical tests. She will document the kind of injury and give him or her rehabilitation and return-to-sport guidelines.

Baseline data of the participants who experienced injury will be correlated with the corresponding data of those who did not, using specific statistical analysis methods to disclose the aetiologic parameters. According to the results, at the next stage, a predictive model for shoulder injury incidence will be created using machine learning. The researchers of the present study aim to generate a model which be able to prognosticate the athletes who are going to be injured in whichever shoulder presenting high accuracy and low overfitting.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults CrossFit participants of any level of experience
* Novices who have already completed the trial workouts

Exclusion Criteria:

* Injured CrossFit participants who have not yet returned to ordinary training

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 150 (anticipated) healthy individuals who participate in CrossFit. They are training in Crossfit affiliated boxes located at 4 different towns in Greece.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2022-09-24 (Actual); Primary Completion 2023-02-12 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
BMI | Baseline assessment
  Weight (kg) and Height (cm) data will be collected to report BMI in kg/m^2
Demographic, general history and shoulder injuries history, activity and experience level | Baseline assessment
  Participant profile will be formed using an especially designed questionnaire, data will be collected regarding the age, upper limb dominance, months of experience, training volume in hours per week, level of competition, warm up and recovery routines adequacy, details of previous injuries and current situation of shoulder functionality.
Core rotation active range of motion | Baseline assessment
  Right and left core rotation will be measured in degrees utilizing a digital goniometer (HALO digital goniometer, HALO Medical Devices) which has affixed on an aluminum stick. Participant will be holding the stick by hands at the level of scapulas spines and starting rotate his or her core to right and then left direction.
Shoulder active range of motion symmetries | Baseline assessment
  Comparative measurements among shoulders. In an upright position, knees forward and flexed as far as it will be needed in order back and lower back to be attached on the wall, participant will move his/her shoulders toward flexion while maintaining the initial position on the wall. When movement will reach the end point of the available range of motion, the researcher will measure the distances between each wrist and the wall using a measuring tape. The distance may be symmetrical otherwise the shoulder of the upper limb with the bigger distance will be documented as deficient.
  Same procedure in the same body position will be followed for external and internal rotation of the shoulders but movements will be performed with 90 degrees of shoulder abduction and 90 degrees of elbow flexion.
Shoulder stabilizers muscle strength | Baseline assessment
  Maximal strength of each shoulder external and internal rotators will be measured in kilograms of resistance utilizing a handheld digital dynamometer, K-Force Muscle Controller, via K-Force Pro application reporting (Kinvent, Montpellier, France)
Lateral differences in muscle strength between shoulders | Baseline assessment
  The percentage of lateral differences in maximal strength of internal and external rotation between shoulders will be measured utilizing a handheld digital dynamometer, K-Force Muscle Controller, via K-Force Pro application reporting (Kinvent, Montpellier, France)
Hip abductors muscle strength | Baseline assessment
  Maximal strength of each hip abductors muscles will be measured in kilograms of resistance with the use of a handheld digital dynamometer, K-Force Muscle Controller, via K-Force application reporting (Kinvent, Montpellier, France)
Lateral differences in hip abductors strength | Baseline assessment
  The percentage of lateral differences in maximal strength of abduction between hips will be measured utilizing a handheld digital dynamometer, K-Force Muscle Controller, via K-Force Pro application reporting (Kinvent, Montpellier, France)
Muscular endurance of shoulder external rotators | Baseline assessment
  Using the aforementioned dynamometer application, participants will be asked to do 3 sets of 30 seconds isometric hold at the 60% of the maximal previously produced strength by external rotators muscles (outcome 5). 5 seconds rest between sets will be used. The percentage of the time, on which participants can produce the requested amount of power, will be recorded. This measurement will reflect the endurance capability of this muscle group for each shoulder. Measurement data will be collected using a handheld digital dynamometer, K-Force Muscle Controller, via K-Force Pro application reporting (Kinvent, Montpellier, France).
Lateral differences in shoulder external rotators endurance | Baseline assessment
  The percentage of lateral differences in external rotation isometric hold between right and left side will be exported from K-Force Pro application reporting.
Shoulder stability | Baseline assessment
  Closed Kinetic Chain Upper Extremity Stability test (CKCUES) will be performed to evaluate shoulder stability.
CrossFit-specific functional parameters (flexibility, stability, power) using an innovative evaluation tool: CrossFit Functional Assessment Battery for Shoulder (CrossFit FABS) | Baseline assessment
  Flexibility, stability and power will be evaluated using an innovative assessment tool which was developed especially for the purpose of the present research. CrossFit FABS (Functional Assessment Battery for Shoulder) is a CrossFit-specific, functional evaluation battery in regard to shoulder injury risks. It is composed of 6 tests which resulted from a wider tool through applied pilot research: deep air squat, shoulder mobility, upper frontal kinetic chain flexibility, overhead squat facing wall, windmill with kettlebell and sots press. Each test is scored from 0 to 3, using a 3-point scoring scale with a maximum total score of 18 points.
Shoulder injury incidents | Up to 12 months
  Any new or aggravated pre-existing shoulder injury that will be responsible for at least 1-day training or game loss or training modification to avoid specific high-impact exercises will be recorded. Also, the whole progression of the recovery until return-to-sport will be monitored.
Shoulder injury characteristics | Up to 12 months
  Injury profile will be formed using an especially designed objective and subjective assessment questionnaire, including present injury history, correlation with performed exercise, symptoms, observation abnormalities and special diagnostic tests for shoulder pain (clinical assessment). Exact kind of injury will be determined by the researcher.
Disability of injured participants | Up to 12 months
  A self-reported questionnaire for shoulder, the SDQ (Shoulder Disability Questionnaire), will be filled by injured participants via interview method by the researcher.
Pain intensity of injured participants | Up to 12 months
  VAS pain scale will be used to determine shoulder pain intensity in injured participants.

SECONDARY OUTCOMES:
Shoulder injury risk factors | After study completion, 2nd year
  Analyzing data of the injured and non-injured participants will reveal possible risk factors for shoulder injuries.
Predictive modeling for shoulder injury incidence in CrossFit | After study completion, 2nd year
  Using machine learning it is aimed to develop a predictive model able to identify the athletes who are going to be injured in their shoulder, ensuring high accuracy and low overfitting.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Patras, Patras, Peloponnese, Greece

REFERENCES:
- [Background] Bullock GS, Mylott J, Hughes T, Nicholson KF, Riley RD, Collins GS. Just How Confident Can We Be in Predicting Sports Injuries? A Systematic Review of the Methodological Conduct and Performance of Existing Musculoskeletal Injury Prediction Models in Sport. Sports Med. 2022 Oct;52(10):2469-2482. doi: 10.1007/s40279-022-01698-9. Epub 2022 Jun 11. PMID 35689749
- [Background] Schwank A, Blazey P, Asker M, Moller M, Hagglund M, Gard S, Skazalski C, Haugsbo Andersson S, Horsley I, Whiteley R, Cools AM, Bizzini M, Ardern CL. 2022 Bern Consensus Statement on Shoulder Injury Prevention, Rehabilitation, and Return to Sport for Athletes at All Participation Levels. J Orthop Sports Phys Ther. 2022 Jan;52(1):11-28. doi: 10.2519/jospt.2022.10952. PMID 34972489
- [Background] Asker M, Brooke HL, Walden M, Tranaeus U, Johansson F, Skillgate E, Holm LW. Risk factors for, and prevention of, shoulder injuries in overhead sports: a systematic review with best-evidence synthesis. Br J Sports Med. 2018 Oct;52(20):1312-1319. doi: 10.1136/bjsports-2017-098254. Epub 2018 Mar 26. PMID 29581141
- [Background] Angel Rodriguez M, Garcia-Calleja P, Terrados N, Crespo I, Del Valle M, Olmedillas H. Injury in CrossFit(R): A Systematic Review of Epidemiology and Risk Factors. Phys Sportsmed. 2022 Feb;50(1):3-10. doi: 10.1080/00913847.2020.1864675. Epub 2021 Jan 7. PMID 33322981
- [Background] Silva ER, Maffulli N, Migliorini F, Santos GM, de Menezes FS, Okubo R. Function, strength, and muscle activation of the shoulder complex in Crossfit practitioners with and without pain: a cross-sectional observational study. J Orthop Surg Res. 2022 Jan 15;17(1):24. doi: 10.1186/s13018-022-02915-x. PMID 35033136
- [Background] Torres-Banduc MA, Jerez-Mayorga D, Moran J, Keogh JWL, Ramirez-Campillo R. Isokinetic force-power profile of the shoulder joint in males participating in CrossFit training and competing at different levels. PeerJ. 2021 Sep 17;9:e11643. doi: 10.7717/peerj.11643. eCollection 2021. PMID 34616590
- [Background] Montalvo AM, Shaefer H, Rodriguez B, Li T, Epnere K, Myer GD. Retrospective Injury Epidemiology and Risk Factors for Injury in CrossFit. J Sports Sci Med. 2017 Mar 1;16(1):53-59. eCollection 2017 Mar. PMID 28344451